CLINICAL TRIAL: NCT06815991
Title: A Phase 1, Single Ascending Dose Administration of MIB-725 to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Community Dwelling Healthy Adults
Brief Title: Phase 1a Single Ascending Dose Study of MIB-725 in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Metro International Biotech, LLC (Industry)
Responsible Party: Principal Investigator, Shalender Bhasin, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIB-725-101
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Healthy Adults
Keywords: Phase 1; NAD Booster

STUDY DESIGN:
Intervention Model Description: This is a single ascending dose study in which 4 different doses of MIB-725 will be administered in ascending order starting with the lowest dose.
Masking Description: Because this is a phase one ascending dose study, masking is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and pharmacokinetic single dose ascending dose study (Experimental): This is a single dose ascending study in which 100, 200, 400, or 800 mg of MIB-725 will be administered as a single oral dose in ascending order starting with the lowest (100 mg) dose
  Interventions: Drug: MIB-725

INTERVENTIONS:
Drug: MIB-725 — MIB-725 is a modified precursor of the NAD+ biosynthetic pathway.

SUMMARY:
This is a single center, open label (i.e. participants and study staff will not be masked to the intervention) single ascending dose study to evaluate the safety, tolerability, pharmaokinetics and pharmacodynamics of MIB-725 in community dwelling, healthy adults. Up to 4 successive groups (cohorts) of 8 subjects each will be enrolled in this trial.

This study will determine the safety and tolerability of orally administered single ascending (increasing) doses (100, 200, 400, and 800 mg) of MIB-725 in healthy adults. The safety will be assessed by evaluating physical examination that includes an external eye examination, vital signs, adverse events, and changes in blood counts, EKG, urinalysis, coagulation measures, and blood chemistries, including but not limited to blood glucose, electrolytes, creatinine, liver function tests, uric acid, and creatine kinase.

DETAILED DESCRIPTION:
Nicotinamide adenine dinucleotide (NAD), a critically important cofactor for the functioning of all living cells, is required for the enzymatic processes that generate energy within the cell, through ATP production during glycolysis, the Krebs cycle, and oxidative phosphorylation (1-3). NAD+ also serves as a co- factor for enzymes, such as the sirtuin and PARP families of enzymes, that modify proteins regulating gene expression, and are involved in DNA repair, inflammation, and innate immune response. Reduced levels of NAD+ are associated with age-related diseases, including metabolic disorders, cancer, and neurodegenerative diseases. Therefore, there is enormous interest in developing therapeutic strategies to raise cellular NAD+ levels with the goal of preventing and treating age-related conditions and diseases in which NAD+ is depleted.

MIB-725 is a modified precursor in the NAD+ biosynthetic pathway. After its oral administration, MIB-725 undergoes biotransformation to produce NAD+. Metro International Biotech is developing this compound for the prevention and treatment of age-related diseases with specific initial focus on the prevention of acute kidney injury (AKI) in at-risk adults who are undergoing coronary artery bypass surgery. Towards this long- term goal, the proposed Phase 1 trial will determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple ascending doses of MIB-725.

This is Phase 1 study of a two part study that will have a separate submission. The first part is an SAD study in which 100, 200, 400, or 800 mg of MIB-725 will be administered as a single oral dose in ascending order starting with the lowest (100 mg) dose. The selection of these doses was informed by the toxicology and pharmacology studies in rats and Beagle dogs. Four groups of participants will be studied. The first group of 8 participants will receive a single dose of 100 mg of MIB-725 orally. If no dose limiting toxicity is observed at this dose, the second cohort (n=8) will receive a single dose of 200 mg MIB-725; the third cohort (n=8) will receive a single dose of 400 mg MIB-725; and the fourth cohort (n=8) will receive a single dose of 800 mg MIB-725. The dose escalation to the next level will be based on the review of the safety data at the lower dose and guided by the pre-specified dose escalation criteria.

The SAD Part 1 will enable the selection of the range of doses and dosing frequencies that can be administered safely in subsequent multiple ascending dose (MAD).

Specific Aims and Objectives Primary Objectives To determine the safety and tolerability of orally administered single ascending doses (100, 200, 400, and 800 mg) of MIB-725 in healthy adults. The safety will be assessed by evaluating physical examination that includes an external eye examination, vital signs, adverse events, and changes in blood counts, EKG, urinalysis, coagulation measures, and blood chemistries, including but not limited to blood glucose, electrolytes, creatinine, liver function tests (ALT, AST, bilirubin, alkaline phosphatase), uric acid, and creatine kinase.

Secondary Objectives To study the pharmacokinetics of orally administered single ascending doses of MIB-725 in healthy adults starting with the 100 mg dose and escalating the dose in ascending order to the maximum dose of 800 mg or a maximal tolerated dose if that is lower than 800 mg.

1. Characterize the time course of blood MIB-725 concentrations and the Caverage 0-24 h concentrations after single administration of each dose level of MIB-725 - 100, 200, 400 and 800 mg.
2. Characterize other single dose PK parameters of MIB-725, such as the observed peak blood concentration (Cmax), time to reach the observed peak blood concentration (Tmax), T1/2 the apparent blood half-life, apparent terminal elimination rate constant, area under the blood concentration versus time curve from time zero to the last measurable concentration (AUClast), area under the blood concentration versus time curve from time zero to 24 hours (AUC24hr), and the area under the blood concentration curve from time zero to infinity (AUCinf) as permitted by the exposure data.
3. Characterize the time course of blood concentrations of metabolites of MIB-725 and their Caverage 0-24 h concentrations after single administration of each dose level of MIB-725 - 100, 200, 400 and 800 mg. Characterize other single dose PK parameters of metabolites of MIB-725, such as the observed peak blood concentration (Cmax), time to reach the observed peak blood concentration (Tmax), T1/2 the apparent blood half-life, apparent terminal elimination rate constant, area under the blood concentration versus time curve from time zero to the last measurable concentration (AUClast), area under the blood concentration versus time curve from time zero to 24 hours (AUC24hr), and the area under the blood concentration curve from time zero to infinity (AUCinf) as permitted by the exposure data.

To characterize the single dose pharmacodynamics of MIB-725 by analyzing the blood concentrations of NAD+, and plasma concentrations of the metabolites of NAD+ and MIB-725. The concentrations in urine of N-methly-2-pyridone-5-carboxamide [2-PY], N-methly-4-pyridone-3-carboxamide [4-PY], nicotinamide, 1-methynicotinamide, nicotinic acid and nicotinuric acid will also be measured.

PK - PD Analyses To relate the changes in MIB-725 dose and circulating concentrations to the change from baseline in blood NAD+ AUC0-24h and plasma concentrations of NAD+-metabolites.

Exploratory Objectives

1. To characterize changes in blood glucose and insulin levels and insulin resistance using HOMA-IR at 2 and 4 hours after a single dose of each of the four dose levels of MIB-725 relative to baseline.
2. To characterize changes in plasma lipids at 24 hours after a single dose of each of the four dose levels of MIB-725 relative to baseline.

Overall Study Design This is a Phase 1 study consisting of 2 parts at a single center (Brigham and Women's Hospital, Boston, MA). This protocol is for part 1 only. Part 1 will be a single dose study in healthy volunteers

General Description of Study Design Single Dose in Healthy Volunteers This is a single center, open label single ascending dose study to evaluate the safety, tolerability, PK and PD of MIB-725 in community dwelling, healthy adults. Up to 4 successive cohorts of 8 subjects each will be enrolled in this trial.

Subjects will be screened for conformity to inclusion and exclusion criteria and those meeting eligibility criteria will be offered participation in the study. Sentinel dosing will be used for the first two dose levels (100 mg and 200 mg). Eight subjects will be enrolled in each cohort to receive a single dose of MIB-725.

MIB-725 will be administered to successive cohorts at escalating dose levels (100, 200, 400 and 800 mg) under fasting conditions. Subjects will be followed for 28 days following dosing according to the Appendix A: Schedule of Events. We will use sentinel dosing for the first two dose levels in. Only one participant will be dosed first with the active drug, and if no severe or serious adverse event is observed in this first participant, the additional participants in that dose cohort will then be dosed at the same dose level. Sentinel dosing will be used in the 100 and 200 mg dose cohorts.

Dose escalation will be sequential and will proceed as long as no pre-defined DLT or stopping criteria are met. Enrollment to the next dose cohort will not commence until an evaluation of all available safety data on all subjects through day 7 of study supports escalation to the next cohort.

Eligible subjects will come to the Clinical Research Unit on Day 1 for approximately 9 hours for administration of the study medication and frequent sampling and observation for 8 hours. After baseline assessments, a single dose of MIB-725 will be administered orally in the Clinical Research Center. Subjects will be discharged after the Hour 8 blood draw and will return for outpatient visits at Hours 24 and 48, and on Days 5, 7, 14 and 28 after study drug administration for evaluations according to the Schedule of Events table.

PK assessments will be performed pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 24, 48, 120, and 168 hours and on day 28 after administration of investigational product.

PD assessments will be performed pre-dose and at specific time points after administration of study drug.

All subjects will be followed for a total of 28 days after investigational product administration.

Estimated Study Duration The study duration for each subject is anticipated to be up to 6 weeks, which includes the screening visit period up to 2 weeks and the 28-day sampling period after investigational product administration. The progression to a higher dose level requires review of the safety data from the entire cohort up to 7 days after the dose by the Safety Review Committee. The 4 dose levels will be studied sequentially. Thus, the trial may take up to 6 months to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Is a non-smoking healthy adult, 19 to 60 years of age, inclusive
2. Has a body mass index (BMI) between 19 and 37.5 kg/m2, inclusive
3. Is free from clinically significant medical problems as determined by the Investigator
4. Is able and willing to provide written informed consent.
5. Is able and willing to provide authorization for the use and disclosure of personal health information in accordance with the Health Insurance Portability and Accountability Act (HIPAA).

Exclusion Criteria:

1. Is a current cigarette smoker
2. AST or ALT > 1.5 times the upper limit of normal
3. Hematocrit < 37% or > 51%
4. Diagnosis of diabetes mellitus, as indicated by use of diabetes medication, hemoglobin A1C > 6.4% or fasting glucose ≥126 mg/dL
5. Serum creatinine > 2.0 mg/dL
6. Current use of barbiturates, benzodiazepines, opiates, amphetamine, cannabinoids and cocaine
7. Known allergy to niacin or nicotinamide mononucleotide
8. Unwilling to refrain from drinking alcohol during the duration of the study
9. Use of any other dietary supplement during the course of the trial
10. Use of anabolic steroids, rhGH, DHEA, androstenedione, or any other performance enhancing drug
11. In the judgment of the study physician, the participant is unlikely to comply with the study protocol for any reason or it may not be safe to administer the study medication
12. Has a history of myocardial infarction, stroke, or heart failure in the preceding 6 months.
13. Has a history of cancer other than nonmelanotic skin cancer requiring treatment in the previous 2 years.
14. Has other medical conditions which, in the opinion of the Principal Investigator, would jeopardize the safety of the study subject or impact the validity of the study results.

In addition, female participants must:

1. Be postmenopausal as indicated by cessation of menstruation at least one year before screening
2. Not be pregnant and not planning to become pregnant over the next 6 months

Prohibited medications and substances:

1. Current use of barbiturates, benzodiazepines, opiates, amphetamine, cannabinoids and cocaine
2. Use of any other dietary supplement during the course of the trial. Subjects who are using a supplement containing nicotinamide, niacin, nicotinamide mononucleotide, or nicotinamide riboside may be included if they agree to stop the supplement at least 2 weeks prior to day 0 and during the entire duration of the study.
3. Initiation of a new prescription drug during the preceding 4 weeks or during the course of the study
4. Use of anabolic steroids, rhGH, DHEA, androstenedione, or any other performance enhancing drug

   -

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events | Baseline to 28 days
  Any treatment-emergent adverse events, including any ocular adverse events
Treatment-emergent serious adverse events | Baseline to 28 days
  Treatment-emergent serious adverse events, including any severe or serious ocular adverse events

SECONDARY OUTCOMES:
Change in blood pressure | Baseline to 28 days
  Change in blood pressure from baseline to 28 days
Change in heart rate | Baseline to 28 days
  Change in heart rate from baseline to 28 days
Presence of conjunctival injection | Baseline to 28 days
  Presence of conjunctival injection during eye examination
Change in QTc interval | Baseline to 28 days
  Change in QTc interval measured using a12-lead electrocardiogram
Pharmacokinetics | Baseline to 28 days
  Blood MIB-725 concentrations measured over time
Pharmacodynamics - blood concentrations of NAD+ levels over time | Baseline to 28 days
  Change in blood concentrations level from baseline to 28 days
Pharmacodynamics - plasma concentrations of NAD+ metabolite,1-methylnicotinamide over time | Baseline to 28 days
  change in plasma concentrations of NAD+ metabolite, 1-methylnicotinamide over time
Pharmacodynamics- plasma concentrations of NAD+ metabolites, 2PY, over time | Baseline to 28 days
  Pharmacodynamics- plasma concentrations of NAD+ metabolites, 2PY, over time
Change in blood concentration of nicotinic acid mononucleotide (NAMN) | Baseline to 28 days
  Change in blood concentration of nicotinic acid mononucleotide (NAMN) from baseline to 28 days
Change in hemoglobin | Baseline to 28 days
  Change in hemoglobin from baseline to 28 days
Change in white blood cell count | Baseline to 28 days
  Change in white blood cell count
Blood chemistry - Change in creatinine | Baseline to 28 days
  Change in creatinine
Blood chemistry - Change in alanine aminotransferase (ALT) | Baseline to 28 days
  Change in ALT
Blood chemistry - Change in asparate aminotransferase (AST) | Baseline to 28 days
  Change in AST

OTHER OUTCOMES:
changes in insulin sensitivity | Baseline to 28 days
  changes in insulin sensitivity measured by the Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Change in total cholesterol | Baseline to 28 days
  Change in total cholesterol
Changes from baseline in triglyceride | Baseline to 28 days
  Change in fasting serum lipid - triglyceride
Change in HDL cholesterol | Baseline to 28 days
  Change in fasting serum lipid: high-density lipoprotein (HDL) cholesterol
Change in LDL cholesterol | Baseline to 28 days
  Change in fasting serum lipid: low-density lipoprotein (LDL) cholesterol
Change in free fatty acids | Baseline to 28 days
  Change in fasting serum lipids - free fatty acids

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MB, BS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No